CLINICAL TRIAL: NCT06979518
Title: A Phase 1, Randomized, Placebo-Controlled, Double-Blind, Parallel-Group Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of GSK3862995B Administered as a Single Dose to Healthy Participants of Chinese, Japanese, and European Ancestry
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of GSK3862995B Administered as a Single Dose to Healthy Participants of Chinese, Japanese, and European Ancestry
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 223982
Record Dates: First submitted 2025-05-13; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: GSK3862995B; Chinese; Japanese; and European ancestry; Healthy Participants; Safety; Tolerability; Pharmacokinetics; Pharmacodynamics; Immunogenicity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: This is a randomized, placebo-controlled, double-blind study
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a double-blind study where participants Care provider (site staff) and investigator will remain blinded throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GSK3862995B (Experimental): Participants of Chinese, Japanese, or European ancestries will receive GSK3862995B.
  Interventions: Drug: GSK3862995B
- Placebo (Experimental): Participants of Chinese, Japanese, or European ancestries will receive matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK3862995B — GSK3862995B will be administered.
  Arms: GSK3862995B
Drug: Placebo — Matching placebo will be administered.
  Arms: Placebo

SUMMARY:
This study aims to assess the ethnic sensitivity of GSK3862995B in terms of safety, tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) in healthy participants of Chinese, Japanese, and European ancestry to enable the inclusion of Chinese and Japanese participants in future global studies.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 50 years of age inclusive
* Participants who are generally healthy as determined by medical evaluation based on screening medical history, physical examination, laboratory tests, and cardiac monitoring
* Body weight of at least 50.0 kilogram (kg) for male participants or at least 45.0 kg for female participants
* Body mass index (BMI) within the range of 18.0 to 28.0 kilogram per square meter (kg/m^2) (inclusive)
* Capable of giving signed informed consent
* Males and females of non-childbearing potential•

Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention or interfering with the interpretation of data
* A history of recurrent infections, or treatment of a chronic infection within 3 months prior to the first dose of study drug
* Abnormal blood pressure (as determined by the investigator)
* Symptomatic herpes zoster within 3 months prior to screening
* Significant allergies to humanized monoclonal antibodies
* Clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe post-treatment hypersensitivity reactions
* Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
* Breast cancer within the past 10 years
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* A clinically significant abnormality in the average of triplicate 12-lead ECG readings performed at screening including
* Antibacterial, antiviral, antifungal, antiparasitic, or antiprotozoal therapy within 30 days of dosing
* Past or intended use of over the counter or prescription medication (including herbal medications) within 7 days prior to dosing and for the duration of study participation
* Live vaccine(s) within 30 days prior to screening or plans to receive such vaccines during the study
* Treatment with biologic agents within 12 weeks, 5 half-lives or twice the duration of the biological effect of the biologic agent (whichever is longer) prior to dosing
* Participation in other clinical study that resulted in loss of blood or blood products >500 millilitres (mL) within a 56 days before participation in this study
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day
* Current enrolment or past participation in another investigational study in which an investigational intervention (e.g., drug, vaccine, invasive device) was administered prior to the first dosing day: 30 days, 5 half-lives, or twice the duration of the biological effect of the investigational product (whichever is longer)
* Current enrolment or past participation in this clinical study
* A positive confirmation of SARS-CoV-2 infection at pre-dose
* Evidence of active or latent Tuberculosis (TB)
* Positive hepatitis Bor hepatitis C test at screening or within 3 months prior to study intervention.
* Positive prestudy drug/alcohol test
* An average weekly intake of >14 units of alcohol
* Regular use of known drugs of abuse, including Tetrahydrocannabinol (THC)
* Current smoker or user or tobacco- or nictotine- containing products, within 30 days prior to screening visit
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study
* Any products intended to treat medical conditions that are not approved by the governing health authority (for example, herbal medicine, health supplements, traditional medicine, homeopathic remedies, etc)
* The participant has a phobia to needles

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2025-11-25 (Estimated); Study Completion 2026-04-27 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AE) | Up to Week 44 (End of follow up visit)
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.
Number of Participants with Serious Adverse Events (SAE) | Up to Week 44 (End of follow up visit)
  An SAE is defined as any untoward medical occurrence that, at any dose, meets one or more of the criteria: results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant, or abnormal pregnancy outcomes (such as, spontaneous abortion, fetal death, stillbirth, congenital anomalies, ectopic pregnancy).
Number of Participants with Clinically Significant Changes in Clinical Laboratory Values | Up to Week 36
  Number of Participants with clinically significant changes in clinical laboratory values (hematology, chemistry and urinalysis) will be assessed.
Number of Participants with Clinically Significant Changes in Vital Signs | Up to Week 36
  Number of Participants with clinically significant changes in vital signs will be assessed.
Number of Participants with Clinically Significant Changes in 12-lead (Electrocardiogram (ECG) | Up to Week 36
  Number of Participants with clinically significant changes in 12-lead ECG will be assessed.
Area Under the Serum Concentration-time Curve Extrapolated to Infinity (AUC[0-inf]) of GSK3862995B | Up to Week 36
  Blood samples will be collected to determine the pharmacokinetic profile of GSK3862995B.
Maximum Observed Concentration (Cmax) of GSK3862995B | Up to Week 36
  Blood samples will be collected to determine the pharmacokinetic profile of GSK3862995B.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/